CLINICAL TRIAL: NCT05251961
Title: The Use Of Growing Rods In Pediatric Long Bones Deformity Correction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelmajeed Aboelabaas Abdelmajeed, principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: pediatric deformity correction
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Deformity of Limb

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: operative deformity correction — * The participants will be subjected to surgical correction using growing rods as a novel technique for their long bone deformities.
  * Procedure will be done under anaesethia
  * Osteotomy , fracture reduction , deformity correction will be done , then introduction of the growing rod

SUMMARY:
The objective of this study is to evaluate the value of growing rods for the correction of long bone deformities in pediatric cases attending Sohag University Hospital and follow up aiming at determining benefits and obstacles to this technique

DETAILED DESCRIPTION:
* The participants will be subjected to surgical correction using growing rods as a novel technique for their long bone deformities.
* Procedure will be done under anaesethia
* Osteotomy , fracture reduction , deformity correction will be done , then introduction of the growing rod

ELIGIBILITY:
Inclusion Criteria:

* cases of osteogenesis imperfecta
* metabolic bone deformities
* cases of hemimelia
* traumatic bone deformities
* complex or simple deformities

Exclusion Criteria:

* adult deformities
* short bone deformities
* very narrow medulla
* osteopetrosis

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The Use Of Growing Rods In Pediatric Long Bones Deformity Correction | 2 years
  - Evaluation of deformity angles correction after use of growing rods in comparison with preoperative angle

REFERENCES:
- [Background] Sarikaya I, Seker A, Erdal OA, Gunay H, Inan M, Guler B. Using a corkscrew-tipped telescopic nail in the treatment of osteogenesis imperfecta: a biomechanical study and preliminary results of 17 consecutive cases. J Pediatr Orthop B. 2019 Mar;28(2):173-178. doi: 10.1097/BPB.0000000000000537. PMID 30216208
- [Background] Persiani P, Ranaldi FM, Martini L, Zambrano A, Celli M, D'Eufemia P, Villani C. Treatment of tibial deformities with the Fassier-Duval telescopic nail and minimally invasive percutaneous osteotomies in patients with osteogenesis imperfecta type III. J Pediatr Orthop B. 2019 Mar;28(2):179-185. doi: 10.1097/BPB.0000000000000536. PMID 30212425